CLINICAL TRIAL: NCT05506566
Title: 68Ga-FAP-CHX PET/CT : Dosimetry and Preliminary Clinical Translational Studies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director of Nuclear Medicine Department, First Affiliated Hospital of Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-FAP-CHX
Record Dates: First submitted 2022-08-14; First posted 2022-08-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Tumor; Positron-Emission Tomography
MeSH Terms: conditions — Neoplasms | interventions — 68Ga-FAPI; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part I: safety, tolerability, biodistribution and dosimetry (Experimental): PET imaging will begin at 30s (30s/bed), 15min (1 min/bed), 30min (2 min/bed), 60min (2 min/bed) and 120min (2 min/bed) after injection, and whole-body low-dose CT needed to be re-acquired at 120 minutes
  Interventions: Drug: 68Ga-FAP-CHX
- Part II: diagnostic efficacy (Experimental): Participants with various types of cancer will have PET imaging 50-100 minutes after injection of 68Ga-FAP-CHX and another agent (68Ga-FAPI-04 or 18F-FDG).
  Interventions: Drug: 68Ga-FAP-CHX

INTERVENTIONS:
Drug: 68Ga-FAP-CHX — The dose will be 0.05 (mCi / kg) +/- 10% given intravenously at a single time prior to imaging
  Arms: Part I: safety, tolerability, biodistribution and dosimetry
Drug: 68Ga-FAP-CHX — 68Ga-FAP-CHX, the dose will be 0.05 (mCi / kg) +/- 10% given intravenously at a single time prior to imaging； 68Ga-FAPI-04, the dose will be 1.8 (MBq / kg) +/- 10% given intravenously at a single time prior to imaging； 18F-FDG, the dose will be 3.7 (MBq / kg) +/- 10% given intravenously at a single time prior to imaging；
  Other Names: 68Ga-FAPI-04; 18F-FDG
  Arms: Part II: diagnostic efficacy

SUMMARY:
As an emerging molecule targeting FAP, 68Ga-FAP-CHX is promising as an excellent imaging agent applicable to various cancers. In this study, we observed the safety, biodistribution and radiation dosimetry of 68Ga-FAP-CHX in patients with various types of cancer and compared them with the results of 68Ga-FAPI-04 or 18F-FDG imaging to evaluate the dosimetric characteristics and diagnostic efficacy of 68Ga-FAP-CHX.

DETAILED DESCRIPTION:
Fibroblast activation protein (FAP) is highly expressed in the stroma of a variety of human cancers and is therefore considered promising for guiding targeted therapy. The recent development of quinoline-based PET tracers that act as FAP inhibitors (FAPIs) demonstrated promising results preclinically and already in a few clinical cases. 68Ga-FAP-CHX is a novel FAP-targeted tracers. The present study aimed to evaluate the biodistribution, pharmacokinetics, and dosimetry of 68Ga-FAP-CHX, and performed a head-to-head comparison with 68Ga-FAPI-04 or 18F-FDG PET/CT scans in patients with various cancers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years < Age < 75 years
* Various solid tumors with available histopathological findings, and have not been treated surgically.
* Signed informed consent.

Exclusion Criteria:

* patients with pregnancy
* the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Human biodistribution | From right after tracer injection to 2-hours post-injection
  reported as relative uptake values per organ at 30s, 15min, 30min, 60min and 120 min per individual subject and as a mean over all subjects (Part I)
Human dosimetry | From right after tracer injection to 2-hours post-injection
  radiation dose to individual organs and the equivalent dose for the whole body of each subject and as a mean over all subjects (Part I). Dosimetry will be calculated using the OLINDA software.
Standard uptake value (SUV) | Up to 2 weeks
  Determination of SUV for detected lesions and discernible organs of 68Ga-FAP-CHX and 68Ga-FAPI-04 or 18F-FDG
Lesion numbers | Up to 2weeks
  Determination of lesion numbers of 68Ga-FAP-CHX and 68Ga-FAPI-04 or 18F-FDG
the sensitivity of 68Ga-FAP-CHX PET/CT | Up to 2 weeks
  compared with pathology or composite imaging, the sensitivity of 68Ga-FAP-CHX PET/CT was evaluated.
the specificity of 68Ga-FAP-CHX PET/CT | Up to 2 weeks
  compared with pathology or composite imaging, the specificity of 68Ga-FAP-CHX PET/CT was evaluated.
the accuracy of 68Ga-FAP-CHX PET/CT | Up to 2 weeks
  compared with pathology or composite imaging, the accuracy of 68Ga-FAP-CHX PET/CT was evaluated.

SECONDARY OUTCOMES:
Count of participants with treatment emergent adverse events | Up to 3 days
  The frequency and severity of treatment emergent adverse events following 68Ga-FAP-CHX injection will be descriptively reported as classified and graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Expression ability of 68Ga-FAP-CHX in different types of tumors | Up to 3 days
  Differentiation of SUVmax in different tumors

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Study Chair — The First Affiliated Hospital, Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No